CLINICAL TRIAL: NCT05331365
Title: Construction and Validation of a Score Evaluating the Residual Instability of the Patient After Ankle Ligamentoplasty - Ankle Go Study
Brief Title: Construction and Validation of a Score Evaluating the Residual Instability of the Patient After Ankle Ligamentoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ankle Go study; 2021-A03239-32 (Other: ANSM)
Record Dates: First submitted 2022-04-04; First posted 2022-04-15 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Ankle Sprains; Ligament Sprain
Keywords: ligamentoplasty; chronic ankle instability; score
MeSH Terms: conditions — Ankle Injuries | interventions — Facility Design and Construction

STUDY DESIGN:
Intervention Model Description: Patients who have undergone ankle ligamentoplasty 4 months ago will be included in the study.
  Healthy volunteers will be selected on a voluntary basis at the request of the investigators in the population of patients undergoing rehabilitation by physiotherapists at the investigation sites and with no history of knee or ankle problems.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group of the construction of the composite Ankle go score and internal validations (Experimental): 50 patients will be include for the construction of the composite score and its internal validations. They will complete questionnaires (FAAM, ALR-RSI) and undergo tests (SLSTS, SHTS, SEBT and Figure of 8) 4 months after ankle's surgery (visit 1), 6 months after surgery (visit 2) and 12 months post surgery
  Interventions: Other: Construction and evaluation of a composite score evaluating post ankle surgery residual instability by completing questionnaires and undergoing physical tests
- group of the external validation stage of the composite score (Experimental): 50 additional patients for the external validation stage of the composite score. They will complete questionnaires (FAAM, ALR-RSI) and undergo tests (SLSTS, SHTS, SEBT and Figure of 8) 4 months after ankle's surgery (visit 1) and 6 months after surgery (visit 2)
  Interventions: Other: Construction and evaluation of a composite score evaluating post ankle surgery residual instability by completing questionnaires and undergoing physical tests
- Group allowing the assessment of the score's ability to discriminate (No Intervention): 30 healthy volunteers (who did not undergone an ankle's surgery) will be included in the study to analyze the ability of composite score to discriminate. The healthy population will perform the same physical and psychological tests as Group allowing the construction of the composite Ankle go score and internal validations

INTERVENTIONS:
Other: Construction and evaluation of a composite score evaluating post ankle surgery residual instability by completing questionnaires and undergoing physical tests — Four tests and two questionnaires, each evaluating specific physical or psychological dimensions will be used to construct the composite score "Ankle Go Test" composite score:
  * Foot and Ankle Ability Measure Questionnaire (FAAM)
  * Ankle ligament reconstruction-return to sport after injury Questionnaire(ALR-RSI)
  * Single Leg Stance Test (SLST)
  * Side Hop Test (SHT)
  * Star Excursion Balance Test (SEBT)
  * Figure-of-8
  Arms: Group of the construction of the composite Ankle go score and internal validations; group of the external validation stage of the composite score

SUMMARY:
The goal of this prospective, open label study is the construction and the evaluation of a composite score evaluating the residual instability in patients who have undergone an ankle's ligamentoplasty (the Ankle Go Test score).

The main hypothesis of this study is based on the fact that the composite score "Ankle Go Test" would allow a global validation of all the criteria of scores of 4 tests and 2 questionnaires, which are performed in common pratice, evaluating the instability of the ankle after an ankle ligamentoplasty.

Participants will have to complete 2 questionnaires (FAAM, ALR RS) and to undergoe 4 tests (Single Leg Stance Test, Side Hop Test, Start Excursion Balance Test, La figure of 8), at 4, 6 and 12 months post surgery.

Researchers will compare the group of participants who undergone ankle's ligamentoplasty with a group of healthy volunteers to assess the discriminant validity of the Ankle Go Test score

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients who underwent arthroscopic ankle ligamentoplasty or healthy volunteers with no previous knee or ankle history.
2. Age ≥ 18 years
3. Patients who's been informed about the study and who didn't express their opposition to participate

Exclusion Criteria:

1. Patients with chronic ankle instability, operated or not, contralateral
2. Patients under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The construction of the " Ankle Go Test ", composed of the scores obtained from the 4 tests and 2 questionnaires perfomed 6 months post ankle's surgery | At 6 months post-intervention
  Three steps will be required to construct the "Ankle Go Test":
  * Determining how much information the tests and questionnaires will contribute to the overall composite score (step 1)
  * Construction of the score itself and extraction of a residual instability cut-off by the patient at 6 months post-intervention (step 2).
  * Confirmation of the weighting and validation of the composite score and the cut-off using an external population (external validation; step 3)

SECONDARY OUTCOMES:
The composite score's sensibility to change (ability of the composite score to measure patients' progress) | At 4 months, 6 months and 1 year post-intervention
  The ability of the composite score to measure patients' progress will be measured by analysis of composite score results at 4 months, 6 months and 1 year post surgery
Reproductibility of the composite score | At 6 months with interval of + 24 hours
  The reproductibility of the composite score will be measured by Analysis of composite score results at 24 hours interval.
Discriminating ability of the composite score | At 6 months post-intervention
  Discriminating ability of the composite score will be measured by the Comparison of the composite score's results in post-operative patients to composite score's results in healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Santé Atlantique, Nantes, France

REFERENCES:
- [Result] Lopes R, Andrieu M, Cordier G, Molinier F, Benoist J, Colin F, Thes A, Elkaim M, Boniface O, Guillo S, Bauer T; French Arthroscopic Society. Arthroscopic treatment of chronic ankle instability: Prospective study of outcomes in 286 patients. Orthop Traumatol Surg Res. 2018 Dec;104(8S):S199-S205. doi: 10.1016/j.otsr.2018.09.005. Epub 2018 Sep 21. PMID 30245066
- [Result] Lopes R, Noailles T, Brulefert K, Geffroy L, Decante C. Anatomic validation of the lateral malleolus as a cutaneous marker for the distal insertion of the calcaneofibular ligament. Knee Surg Sports Traumatol Arthrosc. 2018 Mar;26(3):869-874. doi: 10.1007/s00167-016-4250-7. Epub 2016 Aug 6. PMID 27497693
- [Result] Jure D, Blache Y, Degot M, Vigne G, Nove-Josserand L, Godeneche A, Collotte P, Franger G, Borel F, Rogowski I, Neyton L. The S-STARTS Test: Validation of a Composite Test for the Assessment of Readiness to Return to Sport After Shoulder Stabilization Surgery. Sports Health. 2022 Mar-Apr;14(2):254-261. doi: 10.1177/19417381211004107. Epub 2021 Apr 9. PMID 33834924
- [Result] Blakeney WG, Ouanezar H, Rogowski I, Vigne G, Guen ML, Fayard JM, Thaunat M, Chambat P, Sonnery-Cottet B. Validation of a Composite Test for Assessment of Readiness for Return to Sports After Anterior Cruciate Ligament Reconstruction: The K-STARTS Test. Sports Health. 2018 Nov/Dec;10(6):515-522. doi: 10.1177/1941738118786454. Epub 2018 Jul 19. PMID 30024344
- [Result] Carcia CR, Martin RL, Drouin JM. Validity of the Foot and Ankle Ability Measure in athletes with chronic ankle instability. J Athl Train. 2008 Apr-Jun;43(2):179-83. doi: 10.4085/1062-6050-43.2.179. PMID 18345343
- [Result] Borloz S, Crevoisier X, Deriaz O, Ballabeni P, Martin RL, Luthi F. Evidence for validity and reliability of a French version of the FAAM. BMC Musculoskelet Disord. 2011 Feb 8;12:40. doi: 10.1186/1471-2474-12-40. PMID 21303520
- [Result] Docherty CL, Arnold BL, Gansneder BM, Hurwitz S, Gieck J. Functional-Performance Deficits in Volunteers With Functional Ankle Instability. J Athl Train. 2005 Mar;40(1):30-34. PMID 15902321
- [Result] Franck F, Saithna A, Vieira TD, Pioger C, Vigne G, Le Guen M, Rogowski I, Fayard JM, Thaunat M, Sonnery-Cottet B. Return to Sport Composite Test After Anterior Cruciate Ligament Reconstruction (K-STARTS): Factors Affecting Return to Sport Test Score in a Retrospective Analysis of 676 Patients. Sports Health. 2021 Jul-Aug;13(4):364-372. doi: 10.1177/1941738120978240. Epub 2021 Feb 6. PMID 33550916
- [Result] Gribble PA, Delahunt E, Bleakley C, Caulfield B, Docherty CL, Fourchet F, Fong D, Hertel J, Hiller C, Kaminski TW, McKeon PO, Refshauge KM, van der Wees P, Vicenzino B, Wikstrom EA. Selection criteria for patients with chronic ankle instability in controlled research: a position statement of the International Ankle Consortium. J Orthop Sports Phys Ther. 2013 Aug;43(8):585-91. doi: 10.2519/jospt.2013.0303. Epub 2013 Jul 31. PMID 23902805
- [Result] Martin RL, Irrgang JJ, Burdett RG, Conti SF, Van Swearingen JM. Evidence of validity for the Foot and Ankle Ability Measure (FAAM). Foot Ankle Int. 2005 Nov;26(11):968-83. doi: 10.1177/107110070502601113. PMID 16309613
- [Result] Rosen AB, Needle AR, Ko J. Ability of Functional Performance Tests to Identify Individuals With Chronic Ankle Instability: A Systematic Review With Meta-Analysis. Clin J Sport Med. 2019 Nov;29(6):509-522. doi: 10.1097/JSM.0000000000000535. PMID 31688183
- [Result] Sigonney F, Lopes R, Bouche PA, Kierszbaum E, Moslemi A, Anract P, Stein A, Hardy A. The ankle ligament reconstruction-return to sport after injury (ALR-RSI) is a valid and reproducible scale to quantify psychological readiness before returning to sport after ankle ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2020 Dec;28(12):4003-4010. doi: 10.1007/s00167-020-06020-6. Epub 2020 Apr 30. PMID 32356045